CLINICAL TRIAL: NCT07250815
Title: Infection Outcomes Among Advanced Therapy-naive Older Adult US Patients With UC/CD Initiating ENTYVIO, TNF-alpha Inhibitors, or Ustekinumab: A Retrospective Observational Matched-Cohort Study Using Medicare Claims Data, 2016-2025
Brief Title: A Study on Infections in Adults With Ulcerative Colitis/Crohn's Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Vedolizumab-4081; EUPAS1000000767 (Other: HMA-EMA RWD Catalogue)
Record Dates: First submitted 2025-11-18; First posted 2025-11-26 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Ulcerative Colitis; Crohn's Disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Participants with UC: Participants diagnosed with UC who initiated treatment with ENTYVIO or other advanced medical therapies (AMTs) will be identified using a claims-based algorithm. This algorithm incorporates International Classification of Diseases, 10th Revision, Clinical Modification (ICD-10-CM) codes, National Drug Codes (NDC), and Healthcare Common Procedural Coding System (HCPCS) codes to retrospectively assess the safety outcomes data over a period of approximately four months.
  Interventions: Other: No intervention
- Participants with CD: Participants diagnosed with CD who initiated treatment with ENTYVIO or other AMTs will be identified using a claims-based algorithm. This algorithm incorporates ICD-10-CM codes, NDC, and HCPCS codes to retrospectively assess the safety outcomes data over a period of approximately four months.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is an observational study, no intervention will be administered.

SUMMARY:
More older people (more than 65 years of age) around the world are getting Ulcerative Colitis (UC) or Crohn's Disease (CD). This is happening because people are living longer and because more people overall are developing UC or CD. Medicines that treat UC/CD, however, might make it easier for older adults to get infections.

The main aim of this study is to learn if there is a difference in the number and type of infections in older people when treated with either ENTYVIO or other advance medicines (TNF-alpha inhibitors or ustekinumab) that reduce swelling and pain by blocking a chemical in the body (called TNF-alpha).

The study will include people aged 65 years and older UC or CD who used either ENTYVIO with ustekinumab or a TNF-alpha inhibitor between 2016 and 2025.

Data will be collected from existing Medicare databases.

ELIGIBILITY:
Inclusion Criteria:

UC Study Cohort:

Participants will be included if they had:

-Greater than or equal to (>=) 1 medical (for Medicare fee-for-service [FFS], Part A/B) or pharmacy claim (for Medicare FFS, Medicare Part D) for an approved AMT for UC during the participant identification period.

Note: Claim should be on or after the food and drug administration (FDA) treatment-specific approval dates for each drug.

The date of the first claim during the participant identification period will be designated the Index Date, and the corresponding AMT, the index AMT.

* >=2 medical (for Medicare FFS, Part A/B) claims, at least 30 days apart, with an ICD-10-CM code for UC during the baseline period or on the Index Date.
* Continuous enrollment in either Medicare FFS or Medicare Advantage medical and pharmacy benefits during the Baseline Period.

CD Study Cohort:

Participants will be included if they had:

- >=1 medical (for Medicare FFS, Part A/B) or pharmacy claim (for Medicare FFS, Part D) for an approved AMT for CD during the Participant Identification Period.

Note: Claim should be on or after the FDA treatment-specific approval dates for each drug.

The date of the first claim during the Patient Identification Period will be designated the Index Date, and the corresponding AMT, the index AMT.

* >=2 medical (for Medicare FFS, Part A/B) claims, at least 30 days apart, with an ICD-10-CM code for CD during the Baseline Period or on the Index Date.
* Continuous enrollment in either Medicare FFS or Medicare Advantage medical and pharmacy benefits during the Baseline Period.

If a participant has both a UC and CD diagnosis during the baseline period or on the index date, the diagnosis most proximate to or on the index date will be used to categorize the participant as having UC or CD.

Exclusion Criteria:

Participants with any of the following will be excluded from the analysis:

* Any evidence of AMT utilization during the Baseline Period.
* Participants with at least 2 ICD-10-CM codes for rheumatoid arthritis, ankylosing spondylitis, plaque psoriasis, hidradenitis suppurativa, juvenile idiopathic arthritis, non-infectious uveitis, or psoriatic arthritis during the Baseline Period.
* Participants with 2 or more ICD-10-CM codes for non-dermatologic malignancy during the Baseline Period.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: United States (US) adult participants diagnosed with UC or CD who initiated ENTYVIO or other AMTs will be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 23900 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Hospitalized Due to Serious Infections | Up to 4 months
  Serious infections will include infections of the respiratory tract, skin and soft tissue, genitourinary tract, gastrointestinal tract, central nervous system, and septicemia/sepsis. The intraabdominal infections, perianal infections, tuberculosis, and other opportunistic infections will not be considered under serious infection requiring hospitalization.

SECONDARY OUTCOMES:
Percentage of Participants with Non-serious Infections | Up to 4 months
  Non-serious infections will include any primary diagnosis of infection that is not associated with hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: Click here for more information about this trial in easy-to-understand language, including a Plain Language Summary of the results if the trial has been completed. — https://clinicaltrials.takeda.com/study-detail/8465a8874a244ccf??page=1&idFilter=Vedolizumab-4081